CLINICAL TRIAL: NCT02053922
Title: The Use of Oxytocin, Carbetocin and Buccal Misoprostol in Patients Undergoing Elective Cesarean Section
Brief Title: The Use of Oxytocin, Carbetocin and Buccal Misoprostol in Patients Undergoing Elective Cesarean Section (CS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, karim H abdel-maeboud, Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OCMCS; ASU maternity Hospital (Registry Identifier: ASU maternity Hospital)
Record Dates: First submitted 2013-03-27; First posted 2014-02-04 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Postpartum Hemorrhage
Keywords: caesarean section, ecbolics, postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; carbetocin; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Syntocinon (Active Comparator): Drug is given just after delivery of the neonate during cesarean section.
  Interventions: Drug: Syntocinon
- Carbetocin (Active Comparator): Drug is given just after delivery of the neonate during cesarean section.
  Interventions: Drug: Carbetocin
- Misoprostol (Active Comparator): Drug is given just after delivery of the neonate during cesarean section.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Syntocinon — Syntocinon ampoules (10 IU Oxytocin). (Novartis Pharma, Egypt) One ampoule 10 IU diluted in 10 ml normal saline and administered slowly (over 30- 60 seconds) intravenously just after delivery of the neonate during CS, followed by an intravenous drip of 20 IU oxytocin in 500 ml saline over 4 hours.
  Arms: Syntocinon
Drug: Carbetocin — Carbetocin (Ampoule 100 μg/ml) . [Pabal, Marketing Authorization Holder: Ferring GmbH (Gesellschaft mit beschränkter Haftung), Kiel ,Germany. Manufactured by DRAXIS Pharma , a division of specialty Pharmaceuticals Inc. Montreal ,Canada] ,diluted in 10 ml normal saline and administered slowly (over 30- 60 seconds) intravenously just after delivery of the neonate during CS.
  Other Names: Pabal
  Arms: Carbetocin
Drug: Misoprostol — Misoprostol (200 mcg Tablet) [Misotac, Sigma Pharmaceutical Industries, SAE, Egypt] Two tablets (400 mcg) in the buccal space just after delivery of the neonate during CS.
  Other Names: Misotac
  Arms: Misoprostol

SUMMARY:
The use of Oxytocin, Carbetocin and buccal misoprostol in patients undergoing elective Cesarean Section

DETAILED DESCRIPTION:
The use of Oxytocin, Carbetocin and buccal misoprostol in patients undergoing elective Cesarean Section in the prevention of uterine atony and postpartum hemorrhage (PPH) after caesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Gestational age of pregnancy of 37 completed weeks or more.
3. Written and signed informed consent by the patient to participate in the study.

Exclusion Criteria:

1. fetal or maternal distress where, due to time constraints, it will not possible and/or appropriate to recruit or randomize.
2. Women undergoing caesarean section with general anesthesia are also excluded, because carbetocin is licensed for use with regional anaesthesia only.
3. Women planned to have any other type of uterine incision other than transverse lower segment.
4. Women with HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count), eclampsia, and epilepsy .
5. Women with placental abruption are excluded because there is a higher risk of hemorrhage with this condition and it was therefore felt to be inappropriate to recruit these women.
6. Women with thrombocytopenia, known coagulopathies, or receiving anticoagulant therapy.
7. Women with history of significant heart disease, a history or evidence of liver, renal, vascular disease or endocrine disease (other than gestational diabetes).
8. Women with history of hypersensitivity to oxytocin or carbetocin.
9. Women with any severe allergic condition or severe asthma.
10. Women with any contraindication to receiving prostaglandins, including known hypersensitivity to misoprostol or other prostaglandins (PGs) or glaucoma.
11. Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of buccal misoprostol in the prevention of uterine atony and postpartum hemorrhage (PPH) after caesarean section | an expected average 1 week

SECONDARY OUTCOMES:
Adverse events recorded during the study. | an expected average 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Karim H Abd-El-Maeboud, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Elbohoty AE, Mohammed WE, Sweed M, Bahaa Eldin AM, Nabhan A, Abd-El-Maeboud KH. Randomized controlled trial comparing carbetocin, misoprostol, and oxytocin for the prevention of postpartum hemorrhage following an elective cesarean delivery. Int J Gynaecol Obstet. 2016 Sep;134(3):324-8. doi: 10.1016/j.ijgo.2016.01.025. Epub 2016 May 25. PMID 27350226